CLINICAL TRIAL: NCT03676894
Title: Pilot Single-masked, Randomized, 3-arm Parallel Study Assessing the Tolerability, Safety and Efficacy of Intraurethral/Intravaginal 2940 Nm Er:YAG Laser Treatment for Stress Urinary Incontinence
Brief Title: Intraurethral/Intravaginal 2940 Nm Erbium Laser Treatment for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fotona d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPD16-001-00
Record Dates: First submitted 2018-09-10; First posted 2018-09-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, 3-arm parallel pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham Treatment (Sham Comparator): Sham Fotona SP Dynamis Treatment - minimum energy delivered through sham handpiece.
  Interventions: Device: Sham Fotona SP Dynamis
- Intravaginal Treatment (Active Comparator): Intravaginal Fotona SP Dynamis Treatment - energy delivered intravaginally.
  Interventions: Device: Intravaginal Fotona SP Dynamis
- Intravaginal and intraurethral Treatment (Experimental): Intravaginal and intraurethral Fotona SP Dynamis Treatment Intravaginal Treatment - energy delivered intravaginally and intraurethrally.
  Interventions: Device: Intravaginal Fotona SP Dynamis; Device: Intraurethral Fotona SP Dynamis

INTERVENTIONS:
Device: Sham Fotona SP Dynamis — Female patients with SUI will be treated with non-ablative Er:YAG laser with Fotona SP Dynamis with sham handpiece.
  Arms: Sham Treatment
Device: Intravaginal Fotona SP Dynamis — Female patients with SUI will be treated intravaginaly with non-ablative Er:YAG laser with Fotona SP Dynamis
  Arms: Intravaginal Treatment; Intravaginal and intraurethral Treatment
Device: Intraurethral Fotona SP Dynamis — Female patients with SUI will be treated intraurethraly with non-ablative Er:YAG laser with Fotona SP Dynamis
  Arms: Intravaginal and intraurethral Treatment

SUMMARY:
Primary objective is to assess the tolerability and safety of the intraurethral 2940nm Er:YAG laser technique in combination with intravaginal 2940nm Er:YAG laser method for the treatment of stress urinary incontinence.

DETAILED DESCRIPTION:
This study is a prospective, randomized, 3-arm parallel pilot study. Study subjects will be women currently experiencing female stress urinary incontinence (SUI) and stress-predominant mixed urinary incontinence (SMUI) with a degree of intrinsic sphincter deficiency for a minimum duration of 6 months prior to enrolment. Diagnosis of SUI with a degree of intrinsic sphincter deficiency will be performed using urodynamic and clinical assessment.

Subjects will undergo sham, intravaginal, and the combination of intravaginal and intraurethral treatment with the 2940 nm Er:yttrium aluminum garnet Er:YAG laser at two time points, 4 weeks apart. Primary objective is to assess the tolerability and safety of the intraurethral 2940nm Er:YAG laser technique in combination with intravaginal 2940nm Er:YAG laser method for the treatment of stress urinary incontinence through 6 months follow-up and extend to 12 months follow-up.

Secondary objective is to assess the effectiveness of the intravaginal and combination of intraurethral/intravaginal laser treatments using subjective and objective measures, as well as improvement in quality of life through 6 months follow-up and extend to 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 80 years
* SUI or MUI with predominantly stress symptoms for more than 6 months
* Has failed 2 previous non-invasive therapies for three (3) months each (e.g. behavioural modification, electrical stimulation, pelvic muscle exercise, biofeedback, and/or drug therapy)
* Confirmed SUI through cough stress test or urodynamics
* Has at least one incontinence episode per 24 hour period measured over three days
* Valsalva leak-point pressure (VLPP) ≤100 cm H2O
* Has a baseline 24h pad weight test ≥ 10 gm
* Has maximum cystometric capacity ≥250 mL
* No pelvic surgery within last 6 months (including prolapse repair, subjects who have residual or recurrent SUI following colposuspension or a sling procedure may be included in the study if the procedure was conducted at least 6 months prior to screening /baseline visit)
* Willing to give informed consent and complete the follow up schedule

Exclusion Criteria:

* Active urinary tract or vaginal infection or other active infections of urinary tract or bladder (urethritis, cystitis or vaginitis)
* Has had three (3) or more cultured-proven bacterial urinary tract infection (UTI) in the last 12 months
* Clinical diagnosis of urge incontinence or urge predominant mixed incontinence
* Has detrusor overactivity on urodynamics
* postvoiding residual (PVR) > 100 ml
* Has had previous urethral surgery (i.e. fistula or diverticula)
* Grade 2 or higher Pelvic organ prolapse (POP) or Pelvic organ prolapse grade > 2 as defined by POP-Q and symptomatic
* Suffers from known polyuria (>3l/24h)
* Has a BMI ≤35 kg/m2
* Has unevaluated hematuria
* Has a neurogenic bladder
* Evidence of dysplasia in a Pap smear (done in the last 24 months)
* Tumours of the Urinary tract
* Previous radiation or brachytherapy to treat pelvic cancer
* Has uncontrolled diabetes
* Has active herpes genitalis
* Pregnancy, lactating, or not practicing adequate contraception and/or planning to get pregnant in the next 12 months
* Had a vaginal delivery within 6 months prior to the Screening/Baseline Visit
* Is currently participating in any other clinical trial, or has participated in another clinical trial within 3 months prior to the Screening/Baseline Visit

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 55 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Tolerability of the 2940nm Er:YAG laser technique by VAS pain scale | 18 months
  The tolerability of intra-urethral/intravaginal Er:YAG laser treatment by VAS pain scale during procedure and by monitoring the use of pain relieving medication post treatment. The Visual Analog Scale for Pain (VAS) is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.
The Safety of intra-urethral/intravaginal Er:YAG laser procedure by recording the incidence and severity of complications | 18 months
  The Safety of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women, as assessed by recording the incidence and severity of complications
The Safety of intra-urethral/intravaginal Er:YAG laser procedure by recording the incidence of device related adverse events | 18 months
  The Safety of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women, as assessed by recording the incidence of device related adverse events
The Safety of intra-urethral/intravaginal Er:YAG laser procedure by measure uroflow and post void residual (PVR) | 18 months
  The Safety of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women, as assessed by measure uroflow and post void residual (PVR) 6 months after the 2ed treatment
The Safety of intra-urethral/intravaginal Er:YAG laser procedure by Questionnaire for voiding symptoms (based on IPSS) | 18 months
  The Safety of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women, as assessed by questionnaire for voiding symptoms (based on IPSS)

SECONDARY OUTCOMES:
The effectiveness of the intravaginal and combination of intraurethral/intravaginal laser treatments by recording 3-day voiding diary | 18 months
  The efficacy of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women by recording of improvement in daily number of incontinence episodes via 3-day voiding diary The 3-day voiding diary is a log used to record number of pads used, incontinence episodes, the activity in which the subject was engaged when the incontinence occurred, and micturitions.
The effectiveness of the intravaginal and combination of intraurethral/intravaginal laser treatments by 24-Hour Pad-Weight Test | 18 months
  The 24-Hour Pad-Weight Test will be used to reflect everyday incontinence. This test, standardized by the International Continence Society, correlates well with UI symptoms, and has good reproducibility.
The effectiveness of the intravaginal and combination of intraurethral/intravaginal laser treatments by ICIQ-UI short form questionnaire | 18 months
  The efficacy of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women reduction in SUI as measured by ICIQ-UI short form questionnaire. The ICIQ-UI Short Form Questionnaire provides a brief and robust measure to assess the impact of symptoms of incontinence on quality of life and outcome of treatment.
The effectiveness of the intravaginal and combination of intraurethral/intravaginal laser treatments by recording patient global impression of improvement (PGI-I) | 18 months
  • The efficacy of intra-urethral/intravaginal Er:YAG laser procedure for the treatment of stress urinary incontinence in women by recording patient global impression of improvement (PGI-I). The Patient Global Impression of Improvement (PGI-I) Questionnaire is a global index that may be used to rate the response of a condition to a therapy (transition scale).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University Urology Associates, Toronto, Ontario
  - Exgogenia, Institute of Anti-Aging and Regenerative Medicine, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No